CLINICAL TRIAL: NCT05545397
Title: Sedation Level Estimation Based on Machine Learning of Quantitative Occipital Electroencephalogram Features in Gastroenteroscopy Patients
Brief Title: Sedation Level on Machine Learning With Electroencephalogram in Painless Gastroenteroscopy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Huiwen Zhang
Record Dates: First submitted 2022-08-24; First posted 2022-09-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Gastritis
Keywords: Deep Sedation; Machine learning; EEG characheristics;; Painless gastroscopy
MeSH Terms: conditions — Gastritis | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Eeg characteristics at waking time, EEG characteristics at sedation time, induced dose of propofol, and each additional dose of propofol
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- The propofol group: Patients undergoing painless gastroenteroscopy under general anesthesia
  Interventions: Drug: Propofol; Device: EEG montior

INTERVENTIONS:
Drug: Propofol — And pump propofol at a rate of 600ml/h. The degree of sedation was assessed by the MOAA/S scale until the depth sadation of the patient during the monitor of EEG
Device: EEG montior — And pump propofol at a rate of 600ml/h. The degree of sedation was assessed by the MOAA/S scale until the depth sadation of the patient during the monitor of EEG

SUMMARY:
Painless endoscopy technology can make patients comfortable under anesthesia, but because of the painless inside.The diagnosis and treatment time of endoscopic examination is short, and the transport is fast. Anesthesia related wind such as deep breathing depression and hypoxemia will occurRisks.Eeg depth monitoring can assist anesthesiologists to evaluate the depth of anesthesia and reduce the risk. Artificial intelligence is adopted.There are few reports on the evaluation of anesthesia depth and drug dosage by electroencephalogram (EEG) monitoring in outpatient patients with painless gastroenteroscopy.

DETAILED DESCRIPTION:
1.examination, and establish brainClassification model of electrogram and sedation depth;2. The EEG characteristics, basic information and propofol were administered to all patients.The dose model of propofol painless gastroenteroscopy was established by machine learning to guide anesthesia Drug use;3. Evaluate the time and space complexity of the model, build the model, and assist the anesthesiologist to individualize the patient Chemical, safe and comfortable management.

ELIGIBILITY:
Inclusion Criteria:

1. Painless gastroenteroscopy patients
2. ASA classification is Ⅰ-Ⅱ
3. Patients who are willing to cooperate
4. No schizophrenia,epilepsy and other neurological diseases

Exclusion Criteria:

1. allergic to propofol
2. Patients who are unwilling to cooperate
3. Patients with psychiatric disorders
4. Patients using sedative drugs for a long time
5. Patients with neuropsychiatric disorders
6. Patients with severe heart, liver, kidney and respiratory diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were eligible for this study were monitored by EEG, and propol was pumped at a rate of 600ml/h，MOAA/S was used to evaluate the depth of anesthesia. EEG was labeled, and the amount of propofol was recorded.The MATLAB software was used to analyze the EEG features, establish the classifier and establish the painless gastroenteroscopy of propofol induction dosage prediction model.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram features | during gastroenteroscopy procedure
  Time feature;frequency feature;Entropy
Propofol dosage | during gastroenteroscopy procedure
  from awake to sedation in painless gastroenteroscopy

SECONDARY OUTCOMES:
physiological parameter(blood pressure ) | during gastroenteroscopy procedure
  from awake to sedation in painless gastroenteroscopy with ECG monitor
physiological parameter(heart rate ) | during gastroenteroscopy procedure
  from awake to sedation in painless gastroenteroscopy with ECG monitor
physiological parameter(oxygen saturation ) | during gastroenteroscopy procedure
  from awake to sedation in painless gastroenteroscopy with ECG monitor
time parameter （Arousal times） | during endoscopy
  with monitor and Anesthesiologist's record
success rate of once endoscopy | during endoscopy
  with monitor and Anesthesiologist's record
Incidence of hypoxemia | during endoscopy
  with monitor and Anesthesiologist's record
Endoscopist satisfaction by questionnaire | during endoscopy
  with monitor and Anesthesiologist's record
vasoactive drugs | during endoscopy
  with monitor and Anesthesiologist's record

CONTACTS AND LOCATIONS:
Locations (1):
- Ningxia Medical University Cardiovascular and Cerebrovascular Disease Hospital, Yinchuan, The Ningxia Hui Autonomous Region, China